CLINICAL TRIAL: NCT04760145
Title: EFFECT OF FLOW RESTRICTION ON BONE QUALITY WITHIN A MULTICOMPONENT EXERCISE PROGRAM FOR OLDER WOMEN WITH OSTEOPOROSIS. SINGLE-BLIND CLINICAL TRIAL.
Brief Title: EFFECT OF FLOW RESTRICTION ON BONE QUALITY WITHIN A MULTICOMPONENT EXERCISE PROGRAM FOR OLDER WOMEN WITH OSTEOPOROSIS.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Albert Pérez Bellmunt, Principal Investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CBAS-2021-11Z
Record Dates: First submitted 2021-02-15; First posted 2021-02-18 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases; Exercise
Keywords: Exercise; Osteoporosis; Blood Flow Restriction
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal; Bone Diseases; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Multicomponent exercise with blood flow restriction
  Interventions: Other: Multicomponent Exercise with Blood Flow Restriction
- Control Group (Active Comparator): Multicomponent exercise without blood flow restriction
  Interventions: Other: Multicomponent Exercise without Blood Flow Restriction

INTERVENTIONS:
Other: Multicomponent Exercise with Blood Flow Restriction — * 10 minutes of initial warm-up.
  * 20 minutes of strength exercises.
  * 10 minutes of resistance exercises.
  * 10 minutes of coordination and balance exercises.
  * 5 minutes of flexibility.
  * 5 minutes of return to calm and relaxation.
  All of this multicomponent training will be performed with blood flow restriction.
  Arms: Intervention Group
Other: Multicomponent Exercise without Blood Flow Restriction — * 10 minutes of initial warm-up.
  * 20 minutes of strength exercises.
  * 10 minutes of resistance exercises.
  * 10 minutes of coordination and balance exercises.
  * 5 minutes of flexibility.
  * 5 minutes of return to calm and relaxation.
  All of this multicomponent training will be performed without blood flow restriction.
  Arms: Control Group

SUMMARY:
HYPOTHESIS:

- A multicomponent exercise program where strength exercises are performed with blood flow restriction obtains better values in densitometry and bone mass of osteoporotic patients with respect to the same multicomponent exercise program where strength is worked without flow restriction.

INTERVENTION:

The recruitment of the population will be carried out between July and November 2021, with the collaboration of the Consorci Sanitari de Terrassa (CST), which brings together a hospital center and different primary care centers (CAP). The primary care physicians and rheumatologists of the CST will receive an e-mail from the hospital management, informing them of the study to be carried out so that, if they consider it appropriate, they can inform their patients.

Intervention of the intervention and control group:

Each volunteer will be assigned to an intervention group either to the control group (CG) or experimental group (EG).

The control group and intervention group will receive the same multicomponent exercise program, based on specific literature for being an effective, safe and feasible training for both elderly people {{2091 Bouaziz, Walid 2016;}} {{2092 Fragala,M. S. 2019;}}, with or without frailty {{2093 Cadore, Eduardo L 2014;}} {{2094 Casas-Herrero, Alvaro 2019;}} {{2088 Fernández-García, Ángel Iván 2020;}} and/or with osteoporosis {{2089 Moradell, Ana 2020;}}. The main difference between both groups is that the experimental group (EG) will perform the strength exercises with flow restriction (BFR) while the control group (CG) will not have any restriction.

The periodicity of both groups will be 2 sessions per week, with a duration of 65 minutes per session and the duration of the intervention of 6 months and a follow-up 12 months after the beginning of the intervention (see scheme).

The training will be supervised at all times by a physiotherapist with more than 10 years of experience in multicomponent exercise. The sessions will include both limb and trunk work and will have a clear functional objective, focusing on activities of daily living (ADL). Each session will work on all the basic physical abilities (strength, balance, endurance, flexibility and coordination) and will be divided into:

* 10 minutes of initial warm-up. This is divided into 8 minutes walking on a treadmill or cyclohergometer with an intensity corresponding to 30% of heart rate reserve. Followed by 2 minutes of active mobilizations in both upper and lower extremities.
* 20 minutes of strength exercises. These will be interspersed with the rest of the exercises and will include the different extremities and trunk. During the first month, training will be carried out with loads corresponding to 20% of 1 repetition maximum (RM) and from the second month onwards it will be increased to 30-35% of 1 RM.
* 10 minutes of resistance exercises. These exercises will be interspersed with the rest to make the session much more enjoyable.
* 10 minutes of coordination and balance exercises. These exercises will be interspersed with the rest of the activities.
* 5 minutes of flexibility. These exercises will be performed interspersed with the strength and endurance exercises.
* 5 minutes of return to calm and relaxation. To facilitate the monitoring of the researcher who will apply the intervention, each group will be subdivided into smaller groups (ratio of 5 subjects per researcher).

DETAILED DESCRIPTION:
BACKGROUND

According to the WHO, osteoporosis is a disorder of the skeleton characterized by impaired bone strength, primarily reflecting poor integration of bone density and quality {{2042 NIH Consensus Development Panel on Osteoporosis Prevention, Diagnosis, and Therapy 2001;}}}. There are two types of osteoporosis, the most common is considered primary or idiopathic and includes juvenile, postmenopausal and senile osteoporosis. Secondary osteoporosis is considered to be that in which the deterioration of bone quality is due to different types of systemic diseases or produced by the intake of certain drugs (mainly glucocorticoids, anticoagulants and diuretics) {{2164 Maggi, S 2006;}}. Primary osteoporosis can affect both sexes, but postmenopausal and older women are more vulnerable to this disease because they possess important risk factors such as the same age and estrogen depletion {{2043 Tella, Sri Harsha 2014;}}.

It is estimated that approximately 200 million women worldwide have osteoporosis, approximately 10% of women in their 60s, 20% of women in their 70s, 40% of women in their 80s, and 67% of women in their 90s {{2044 Kanis, John Anthony 2007;}}}. Double beam X-ray densitometry (DEXA) is the test to accurately determine bone mass {{2046 Curiel, M Diaz 1997;}}{{2045 Peris,P. 2000;}} and osteoporosis is considered to be present when densitometry values are below 2.5 standard deviations (SD) of peak bone mass {{2081 Kanis, John A 1994;}}, the maximum value reached in young women.

The reduced mass and altered microstructure of osteoporotic bone leads to increased bone fragility and an increased risk of bone fracture {{2047 Anonymous 1993;}} {{2048 Norohna, Judith A 2020;}}. It is estimated that an osteoporotic fracture occurs every 3 seconds and 8.9 million such fractures are considered to occur worldwide {{2049 Ribagin, Simeon 2016;}}, accounting in the European continent for 1.75% of noncommunicable diseases {{2051 Johnell, Olof 2006;}}. Fragility fractures are estimated to be associated with significant morbidity and mortality. Johnell and Kanis estimated that 740,000 deaths per year are associated with hip fracture due to osteoporosis {{2052 Johnell, Olof 2004;}}}. Despite advances in therapeutic procedures only 30-45% of those who survive a hip fracture recover pre-fracture function and 32-80% suffer some form of dysfunction {{2142 Rey-Rodriguez,M.M. 2020;}}} {{2144 Takahashi, Ai 2020;}}, thus representing a high economic and life cost for the countries that suffer from them. It is estimated that in 2050 the United States will spend $131.5 billion to treat fractures caused by osteoporosis {{2053 Burge, Russel 2007;}}}.

Associated with osteoporosis, numerous investigations, have observed a correlation between altered bone quality ( osteopenia or osteoporosis) and a decrease in strength and/or muscle mass (sarcopenia) thus increasing the frailty and deterioration of the patient suffering from it {{2054 Hirschfeld, HP 2017;}} {{2055 Hassan, Ebrahim Bani 2017;}} {{2056 Paintin, James 2018;}} {{2056 Paintin, James 2018;}}. Tokeshi et al. observed how patients with osteoporotic fracture had lower muscle mass compared to those patients without osteoporisis {{2057 Tokeshi, Soichiro 2020;}}}. Hoo Lee and Sik Gong describe that lower extremity muscle mass and loss of grip are closely related to the occurrence of osteoporotic vertebral fracture {{2058 Eguchi, Yawara 2019; }} and numerous investigations show the relationship between grip strength and osteoporotic fractures in older elderly {{2059 Kärkkäinen, M 2008;}} {{2060 Denk, Katharina 2018;}} {{2061 Kamiya, Kuniyasu 2019;}} {{2062 Samelson, Elizabeth J 2006;}} {{2062 Samelson, Elizabeth J 2006;}}.

Because of the morbidity, increased associated frailty, and high economic cost associated with osteoporosis, different therapeutic strategies have been proposed. Although the number of patients treated with pharmacology has been increasing in recent years {{2166 de Felipe,R. 2010;}} and treatment recommended in most clinical guidelines {{2167 Sanfélix-Genovés, José 2014;}}{{2165 Tarantino 2017;}}, more global approaches such as exercise and/or nutrition are increasingly gaining importance {{2165 Tarantino 2017;}} {{2168 Jang,H.D. 2020;}}

HYPOTHESIS:

- A multicomponent exercise program where strength exercises are performed with blood flow restriction obtains better values in densitometry and bone mass of osteoporotic patients with respect to the same multicomponent exercise program where strength is worked without flow restriction.

INTERVENTION:

The recruitment of the population will be carried out between July and November 2021, with the collaboration of the Consorci Sanitari de Terrassa (CST), which brings together a hospital center and different primary care centers (CAP). The primary care physicians and rheumatologists of the CST will receive an e-mail from the hospital management, informing them of the study to be carried out so that, if they consider it appropriate, they can inform their patients.

Intervention of the intervention and control group:

Each volunteer will be assigned to an intervention group either to the control group (CG) or experimental group (EG).

The control group and intervention group will receive the same multicomponent exercise program, based on specific literature for being an effective, safe and feasible training for both elderly people {{2091 Bouaziz, Walid 2016;}} {{2092 Fragala,M. S. 2019;}}, with or without frailty {{2093 Cadore, Eduardo L 2014;}} {{2094 Casas-Herrero, Alvaro 2019;}} {{2088 Fernández-García, Ángel Iván 2020;}} and/or with osteoporosis {{2089 Moradell, Ana 2020;}}. The main difference between both groups is that the experimental group (EG) will perform the strength exercises with flow restriction (BFR) while the control group (CG) will not have any restriction.

The periodicity of both groups will be 2 sessions per week, with a duration of 65 minutes per session and the duration of the intervention of 6 months and a follow-up 12 months after the beginning of the intervention (see scheme).

The training will be supervised at all times by a physiotherapist with more than 10 years of experience in multicomponent exercise. The sessions will include both limb and trunk work and will have a clear functional objective, focusing on activities of daily living (ADL). Each session will work on all the basic physical abilities (strength, balance, endurance, flexibility and coordination) and will be divided into:

* 10 minutes of initial warm-up. This is divided into 8 minutes walking on a treadmill or cyclohergometer with an intensity corresponding to 30% of heart rate reserve. Followed by 2 minutes of active mobilizations in both upper and lower extremities.
* 20 minutes of strength exercises. These will be interspersed with the rest of the exercises and will include the different extremities and trunk. During the first month, training will be carried out with loads corresponding to 20% of 1 repetition maximum (RM) and from the second month onwards it will be increased to 30-35% of 1 RM.
* 10 minutes of resistance exercises. These exercises will be interspersed with the rest to make the session much more enjoyable.
* 10 minutes of coordination and balance exercises. These exercises will be interspersed with the rest of the activities.
* 5 minutes of flexibility. These exercises will be performed interspersed with the strength and endurance exercises.
* 5 minutes of return to calm and relaxation. To facilitate the monitoring of the researcher who will apply the intervention, each group will be subdivided into smaller groups (ratio of 5 subjects per researcher).

ELIGIBILITY:
Inclusion Criteria:

* A woman between 60 and 75 years of age with a medical diagnosis of osteoporosis by means of a femur or lumbar densitometry of less than 2.5 standard deviations (SD) of peak bone mass.
* No history of previous fracture in the last 10 years.

Exclusion Criteria:

* Secondary osteoporosis.
* Having suffered a bone fracture in the last year.
* Present primary osteoporosis but who presented juvenile osteoporosis in adolescence or youth.
* Uncontrolled arterial hypertension.
* Severe acute respiratory failure.
* Uncontrolled orthostatic hypotension.
* Diabetes mellitus with acute decompensation or uncontrolled hypoglycemia.
* Endocrine, hematological and other associated rheumatic diseases.
* Mental health problems (schizophrenia, dementia, depression, etc.) or not being in full mental capacity.
* Patients with pharmacological treatments of glucocorticoids, anticoagulants and/or diuretics.
* Patients with coagulation problems or previous cardiac pathology.
* People with a body mass index (BMI) equal to or higher than 30.
* Subjects who present a systemic disease or any other pathology in which therapeutic exercise could be contraindicated.

Ages: 60 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — postmenopausal women
Enrollment: 94 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Dual-energy X-ray absorptiometry (DEXA) | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  s a test that measures the density of your bones. The DEXA scan is an x-ray scan that uses a small amount of radiation to take pictures of different bones. These pictures are used to measure the density of the bones at the spine and hip in this case.
Quantitative Ultrasound (QUS) | Change between baseline(immediately before intervention) and 2, 4, 6 (post intervention), 8, 10 and 12 (final of the study) months after baseline
  is a relatively recent and noninvasive method of estimating bone mineral status at peripheral skeleton. In addition to bone density, QUS methods provide some structural information, which may be important in determining the fracture risk
Osteoporosis self efficacy scale (OSES) | Change between baseline(immediately before intervention) and 2, 4, 6 (post intervention), 8, 10 and 12 (final of the study) months after baseline
  o measure confidence for adopting behavior change regarding calcium intake (6 items) and exercise (6 items).
  Participants are asked, "If it were recommended that you do any of the following THIS WEEK, how confident or certain would you be that you could:" and then presented with a list of examples such as: "Do exercises even if they are difficult" and "Obtain foods that give an adequate amount of calcium even when they are not readily available." Participants then respond on a 10-point Likert-type scale of 0 to 10 (0=not confident at all, 10=very confident). For each participant, an Exercise Score is calculated by averaging the responses to the 6 exercise-related items and multiplying by 10, and a Calcium Score is derived by averaging the responses to the 6 calcium-related items and multiplying by 10 (range: 0-100). Cronbach's alpha coefficients ranged from 0.90 to 0.94

SECONDARY OUTCOMES:
Senior Fitness Test | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The battery includes tests for lower and upper body strength, agility/dynamic balance, lower and upper body flexibility, and aerobic endurance. ... Objective We examined the effect of silent myocardial ischemia (SMI) on functional fitness levels and physical independence
EUROFIT Fitness test battery | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  is a set of nine physical fitness tests covering flexibility, speed, endurance and strength
Physical Activity Scale for the Elderly (PASE) | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  s an easily administered and scored instrument that measures the level of physical activity in individuals aged 65 years and older. The development of this instrument was supported by a Small Business Innovation Research grant from the National Institute on Aging.
Elderly EXERNET Physical Activity Questionnaire (EEPAQ) | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  includes three questions about the time spent sitting, walking and doing household activities per day
6-min-walk test | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The 6 Minute Walk Test is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Chair stand test | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  n which participants stand up repeatedly from a chair for 30 seconds. This test is part of the Senior Fitness Test Protocol, and is designed to test the functional fitness of seniors.
Isometric Power (with MicroFet 2) | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  Assessment of maximal isometric strength of the limbs in kgs.
Flamingo test | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The Flamingo Balance Test is total body balance test, and forms part of the Eurofit Testing Battery. This single leg balance test assesses the strength of the leg, pelvic, and trunk muscle as well as dynamic balance.
Frail Scale | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The FRAIL scale includes 5 components: Fatigue, Resistance, Ambulation, Illness, and Loss of weight (10). Frail scale scores range from 0-5 (i.e., 1 point for each component; 0=best to 5=worst) and represent frail (3-5), pre-frail (1-2), and robust (0) health status
SF-36 questionnaire | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The SF-36 Health Questionnaire is composed of 36 questions (items) that assess both positive and negative health states. The 36 items of the instrument cover the following scales: Physical Function, Physical Role, Bodily Pain, General Health, Vitality, Social Function, Emotional Role, and Mental Health. Additionally, the SF-36 includes a transition item that asks about change in general health status from the previous year. The items are coded, aggregated and transformed into a scale ranging from 0 (worst health status for that dimension) to 100 (best health status).
minimental Test | Change between baseline(immediately before intervention) and post intervention (6 months after baseline); Change between baseline and final of the study (12 months after baseline)
  The Mini-Mental State Exam (MMSE) is a widely used test of cognitive function among the elderly; it includes tests of orientation, attention, memory, language and visual-spatial skills.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos López-de-Celis, PhD, Study Chair — Universitat Internacional de Catalunya